CLINICAL TRIAL: NCT06724354
Title: The Effect of Use of Infection Control Precaution Package on the Rate of SSI in Patients Undergoing Craniotomy
Brief Title: The Effect of Bundle Application on Surgical Site Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Birgül Belgin, nursing, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CukurovaU-HEKK-BB-01
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Craniotomy Surgery; Preventive Health Care
Keywords: Care package,; surgical site infection; infection rate; healthcare associated infection
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection | interventions — Postoperative Period

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled intervention study to investigate the effect of the care bundle application on surgical site infection rate in cranial brain surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The patients in the experimental group were applied a care package protocol. Before the surgery; ensuring that the patient takes a shower, the necessity of shaving, the application of appropriate surgical prophylaxis, and the provision of preoperative glycemic control were applied to the experimental group. During the surgery; ensuring appropriate surgical hand hygiene, complying with aseptic technique, preparing the skin with appropriate antiseptic solution, keeping the patient's body temperature above 36°C during the surgery, repeating antibiotic prophylaxis in prolonged surgeries, and ensuring optimum oxygenation were applied. After the surgery; ensuring aseptic technique during dressing, ensuring hand hygiene before and after each intervention to the wound, not opening the wound for the first 48 hours, not continuing surgical antibiotic prophylaxis for more than 24 hours after the surgery, and the provision of postoperative glycemic control were applied.
  Interventions: Other: The Surgical Site Infections Precaution Package Form includes the parameters that should be applied to patients before, during and after surgery.
- control group (No Intervention): The infection prevention package parameters were not applied and the routine practice of the clinic was continued.

INTERVENTIONS:
Other: The Surgical Site Infections Precaution Package Form includes the parameters that should be applied to patients before, during and after surgery. — Surgical site infections are a preventable cause of morbidity following surgical procedures. Strategies to reduce SSI rates should address preoperative, perioperative and postoperative factors, and multiple interventions can be combined into 'bundles'. Adoption of these measures may reduce SSIs, but this is dependent on a high level of package compliance. The aim of this study was to evaluate the change in SSI rates after the implementation of the SSI prevention package after neurosurgical operations. It is thought that if the results of our study are positive, the package form created will be pioneered for use in other patient groups. In addition, reducing SSI rates will shorten the postoperative recovery time of patients and reduce hospital costs.
  Arms: intervention group

SUMMARY:
Surgical site infections (SSI) are the most common complications after surgical operations and are in the top three in Healthcare Associated Infections (HIE). Due to surgical site infections, morbidity, mortality and hospital stay in postoperative patients increase, as well as the cost of treatment. The World Health Organization (WHO) has published a list of infection control measures, including preoperative, intraoperative and postoperative precautions, in the guideline for the prevention of SSI.

The aim of infection control is to minimize preventable risks. It is recommended to use evidence-based practices for this purpose. Care packages consisting of combining and using high-evidence applications are applications that can benefit the patient. When these applications are done individually, they benefit the patient, but applying them all in the same package gives better results. In the care given using the care package, the health team creates a common language. The fact that these applications are evidence-based provides the opportunity to control patient care, while reducing the cost and complications.

Despite advances in healthcare, SSI is still one of the major causes of morbidity and mortality. Although perioperative infection prevention packages are frequently applied in fields such as general surgery and orthopedic surgery, there are few studies stated that they are applied in neurosurgery operations where the defense mechanism against microorganisms is very low. However, SSI seen after cranial surgery may also cause an increase in morbidity and mortality. It is aimed to reduce CAE with the increasing use of package applications in developed and developing countries in recent years, and it is seen that positive results have been obtained from the studies on package application. However, when the domestic literature was searched, no study on the subject was found. It is thought that the planned study will contribute to the literature in terms of supporting the perioperative recovery of the measures taken to reduce the infection rate.

DETAILED DESCRIPTION:
Healthcare-Associated Infections (HAI) pose a risk to patient safety all over the world and in our country, and cause financial loss by increasing mortality and morbidity rates. Surgical site infections (SSI) constitute approximately 15% to 30% of HAI and are in the top three of these infections. SSI are infections that develop in the relevant incision site, organ or space after a surgery. According to the guide published by the Centers for Disease Control and Prevention (CDC) in 2017, SSI is divided into three categories: superficial incisional, deep incisional and organ/space. Superficial incisional SSI is defined as infections related to the surgical incision and the opened or manipulated area observed within 30 days following the surgical intervention, while deep incisional and organ/space SSI is defined as infections related to the surgical incision and the opened or manipulated area observed within 30 or 90 days following the surgical intervention.

In Europe, SSI has been found to affect more than 500,000 people per year and cost 19 million euros, while in the United States, it causes patients to spend 400,000 extra days in the hospital, costing 10 billion US dollars per year. Infection rates vary by country and type of surgical procedure: SSI occurs in about 2% of the estimated 80 million surgeries performed annually in the United States. In Europe, rates range from 0.6% to 9.5%. A study in Brazil found a surgical site infection rate of 3.4%. A study in 16 provinces in Turkey reported a rate of 4.5%. SSI rates range from 0.9% in the United States, 2.6% in Italy, 2.8% in Australia, and 2.1% in the Republic of Korea.

SSI is a significant health problem in terms of increasing the length of hospital stay and costs. Infection can cause pain, discomfort, loss of income and reduced quality of life for patients. These infections can range from a simple incision site abscess with purulent discharge to a complex infection that can cause a life-threatening situation and possible morbidity.

Measures to reduce infections are necessary to reduce patient morbidity as well as hospital costs and resource use. There are various strategies to prevent infections. The greatest impact has been found in combining different measures in a care package. Care packages, a new approach used to improve patient outcomes, were first defined in 2001 by the Institute for Healthcare Improvement (IHI) to improve clinical outcomes in intensive care patients. Care packages, which are reported to be effective in improving patient outcomes, require the implementation of scientifically proven interventions as a package. If one of the practices in the package is not followed, the other practices are considered not to have been implemented. Due to this feature, the care package is also known as the "all or nothing" standard and is used by creating checklists with "yes" and "no" steps.

Neurosurgery patients are susceptible to infections during and after surgery. In neurosurgical procedures, physical and mechanical barriers that serve as defense mechanisms against microorganisms are disrupted. These patients often carry the risk of multiple hospital-acquired infections due to risk factors such as multiple trauma, head trauma, neurological deficits, coma, and immobilization. Meningitis infections, which are generally considered to be a small proportion of hospital infections, are quite common among SSI infections in cranial surgery. This situation prolongs the length of hospital stay, increases treatment costs, and mortality. Infections after cranial brain surgery are seen in 0.5%-7.2% of patients and cause repeat surgeries, prolonged antibiotic treatment, and increased hospital stay, and are often life-threatening.

In a meta-analysis of 21 studies conducted between 2000 and 2020 to evaluate the incidence of cranial surgical site infections, it was concluded that bundled applications were effective in reducing SSI rates. In a study conducted in a tertiary hospital to evaluate surgical site infection after neurosurgical operations and the effect of the infection prevention package, 322 patients were evaluated before and after the bundle application. It was observed that infection rates decreased from 7.8% to 3.7% 1 year after the bundle application.

The aim of the study is to examine the effect of care package application on surgical site infection rate in cranial surgery. In recent years, package applications have increased in the world and it is aimed to reduce the SSI rate and many studies are being conducted on this subject. In our country, package applications aimed at preventing invasive device-related infections continue, but the application aimed at preventing SSI has not yet been fully implemented. The reasons for this include the lack of a standard SSI prevention package created by the Ministry of Health, the long surgical process and the necessity of working with a multidisciplinary team to ensure package compliance, and many factors such as operating rooms being busy and stressful environments. In this context, it is thought that our study will contribute to the creation of literature on the effect of SSI prevention care package applications on the infection rate in our country and that the measures will reduce the SSI rate.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 18, Those who have had craniotomy surgery, Those who do not have a diagnosed psychiatric disease, Those who have had elective surgery, Those who have had surgery for the first time

Exclusion Criteria:

* Those who underwent emergency surgery, Those who were pregnant, Those who had a foreign object inserted during surgery, Those who had an infection during hospitalization, Those who underwent surgery for the second time with the same surgery code, Those who refused to participate in the study by themselves or their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection rate | 30 days
  The Surgical Site Infection Prevention Care Package applied after cranial surgery has an effect on the rate of SSI development.

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Birgül, Principal Investigator — Cukurova University Health Application and Research Center Balcali Hospital; Erden Sevilay, Study Director — Cukurova University Faculty of Health Sciences Department of Surgical Diseases
Locations (1):
- Cukurova University Health Application and Research Center Balcali Hospital, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No